CLINICAL TRIAL: NCT01702896
Title: Phase II Trial of Moderate Dose Bolus Interleukin-2 in Metastatic Melanoma
Brief Title: Interleukin-2 in Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Decision
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-07
Record Dates: First submitted 2012-10-04; First posted 2012-10-10 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Melanoma Metastatic
Keywords: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interleukin-2 (Experimental): Interleukin-2 will be used in this group
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — Interleukin-2
  Other Names: IL2

SUMMARY:
To determine whether Interleukin-2 at the dose and schedule will help to increase tumor shrinkage

DETAILED DESCRIPTION:
In this phase II trial, the previously described IL-2 schedule (daily IL-2 for 5 days (per week) every 3 weeks) will be tested in a larger cohort of patients with melanoma to attempt to determine the response rate, median duration of response, and median survival. The dose intensity of this schedule would allow a patient treated on this regimen to achieve the target threshold (> 1440 million IU/m2/year).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologic diagnosis of metastatic melanoma. Patients may have received prior systemic therapy or may be previously untreated.
2. Patients must have bi-dimensional measurable disease on physical exam or radiologic studies.
3. ECOG performance status of 0 or 1 and estimated survival of at least 3 months.
4. White blood count of > 3500/mm3, platelet count > 100,000/mm3, hemoglobin > 9.0 gm/dl; bilirubin, ALT, AST < 3 x upper limit of normal; serum creatinine < 2.0 mg/dl.
5. Patients must undergo a low-level cardiac stress test as a screen for possible atherosclerotic heart disease. Patients with a positive stress test would be excluded from this trial.
6. Patients with elevated temperatures > 100.5 F must have sources of occult infection excluded.
7. Patients must be felt to have recovered from effects of prior therapy, such as > 2 weeks after prior chemotherapy.
8. Patient consent must be obtained prior to entrance onto study.
9. Women of childbearing potential must have a negative pregnancy test and must take adequate precautions to prevent pregnancy during treatment

Exclusion Criteria:

1. Medical illness requiring corticosteroids or other immunosuppressive agents (such as cyclosporin or methotrexate.
2. Autoimmune disease such as inflammatory arthritis which could be exacerbated by immune-based therapy.
3. Prior history of psychiatric disorder which could be exacerbated by interleukin-2.
4. Lactation or pregnancy.
5. Evidence of significant cardiovascular disease including history of recent (< 6 months prior) myocardial infarction, congestive heart failure, primary cardiac arrhythmias (not due to electrolyte disorder or drug toxicity, for example) beyond occasional PVC's, angina, positive low-level stress test, or cerebrovascular accident.
6. Current brain metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Waypa, FNP, Study Director — Research Director
Locations (1):
- Western Regional Medical Center, Inc., Goodyear, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Interleukin-2: All patients received Interleukin-2
Period: Overall Study
Arm/Group | Interleukin-2
Started | 8
Completed | 0
Not Completed | 8

BASELINE CHARACTERISTICS:
Groups:
- Number of Participants: Treated with Interleukin-2
Arm/Group | Number of Participants
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Radiographic studies to evaluate for response were done after every 2 cycles (6 weeks) until disease progression or death from any cause up to 2 years. Standard RECIST response criteria were utilized. Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response Rate (ORR) = 100%(CR + PR/total number of patients receiving Interleukin-2).
Time Frame: Measured until Disease Progression or death from any cause up to 2 years
Population: Data not collected
Groups:
- Response Rate: Percentage of patient who received IL-2 that had a positive response to treatment.
Arm/Group | Response Rate
Number analyzed (Participants) | 0

2. Secondary Outcome: Median Duration of Response
Description: Duration of response is calculated as the time (months) from the date at which response is first observed (per standard Response Evaluation Criteria In Solid Tumors [RECIST] to the date of first observed disease progression or date of death from any cause, whichever came first, assessed up to 2 years. The actual date of tumor assessments was used for this calculation. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of one or more new lesions.
Time Frame: Measured until Disease Progression or death from any cause up to 2 years
Population: Data not collected
Arm/Group | Interleukin-2
Number analyzed (Participants) | 0

3. Secondary Outcome: Median Survival
Description: Measured from date of entry on study until date of death
Time Frame: From time of study entry until death, up to 10 years
Population: Data was not collected
Groups:
- Median Survival: Median survival was measured from date of entry on study until date of death
Arm/Group | Median Survival
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Adverse Events: Patients receiving Interleukin-2
Arm/Group | Adverse Events
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes